CLINICAL TRIAL: NCT06175403
Title: Niacin Regulation of Regional Adipose Tissue Lipolysis
Brief Title: A Study of Niacin Regulation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-003673; 2R01DK040484-35A1 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Excessive Weight Gain
MeSH Terms: interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Upper body obesity (Experimental): Subjects identify with upper body obesity will receive Niacin to lean how fat cells in different regions of the body the response.
  Interventions: Drug: Niacin
- Normal weight (Experimental): Subjects identify with normal body weight will receive Niacin to lean how fat cells in different regions of the body the response.
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Niacin — Intravenous administration of dose titrated from 10 µg·kg FFM-1·min-1 to 30 µg·kg for approximately 4.5 hours on one occasion

SUMMARY:
Adults who gain most of their excess weight in the abdominal area typically do not respond to things that "turn off" fat cells the same way as lean people. The researchers are trying to understand why fat tissue responds differently in people with different body types.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age who are able to comprehend instructions, follow study procedures, willing to sign an informed consent form, and consume an isoenergetic diet eating all meals from Mayo CRTU for at least 3 days prior to study.
* Overweight/Obese volunteers will have a BMI 29.0 - 40.0 kg/m2.
* Upper body/visceral obesity (UBO) in women will be defined as those with a waist-hip ratio (WHR) > 0.85 and/or increased visceral fat by single slice CT scan, usually with > 120 cm2 of visceral fat by CT scanning or a visceral fat/total fat ratio of > 0.30, and/or biochemical evidence of metabolic syndrome as defined by ATP III criteria (fasting plasma triglycerides ≥ 150 mg/dL, HDL-cholesterol < 50 mg/dL for women and < 40 mg/dL for men, fasting plasma glucose ≥ 100 mg/dL). Upper body obesity in men will be defined as a waist-hip ratio of > 0.95 and/or increased visceral fat (visceral fat area > 180 cm2 or a visceral/total fat abdominal ratio by CT of > 0.40) by single slice CT scan and/or biochemical evidence of metabolic syndrome as defined by ATP III criterial. These visceral fat values are based upon the data collected at Mayo Clinic using our methods, and are correlated with dyslipidemia and hyperinsulinemia.
* Female subjects are eligible if they meet the following criteria: are not pregnant or nursing; all women of childbearing potential will have a negative urine pregnancy test at screening and a negative urine pregnancy test within 48 hours before administering study drug; all women of childbearing potential will use an appropriate contraceptive method, including barrier method, oral contraceptive medication, contraceptive device or abstinence while participating in the study. They will confirm use of one of these methods.
* Recent or current research participation in a study that involves an investigational drug. Participants in other clinical trials that involve an investigational drug will not be able to participate in this study until 12 weeks after their participation in the other study is complete or > than five half-lives of the compound, whichever is longer: if Yes look at consent form and f/u visits: current use of medications that alter fatty acid or adipose metabolism possibly given: if yes, exclude;
* Amount of blood drawn during the study (if our study plus this one draw ≥ 450 ml these should be separated by 8 weeks.
* Previous labs: HbA1C < 6.5% for non-diabetic UBO; Fasting glucose < 126 mg/dl for non-diabetic UBO; Hb ≥ 11.0 for women and ≥ 12 for men; platelets > 100 000.

Exclusion Criteria:

* Individuals with a history of a disease process such as: ischemic heart disease; atherosclerotic valvular disease; persistent blood pressure greater than 160/95 despite antihypertensive medication.
* Smokers.
* Concomitant use of medications that can alter free fatty acid metabolism: high dose fish oil (>3g per day), (if yes, discontinue for 6 weeks); statins (if yes hold for 4 weeks and receive primary care provider's approval); Niacin; Fibrates; thiazolidinediones; Beta-blockers; Oral or injected corticosteroids or anabolic steroids; any history of use of pioglitazone; atypical antipsychotics.
* Allergy to lidocaine.
* Allergy to Niaspan documented by immunological testing.
* Allergy to indocyanine green.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma free fatty acid (FFA) concentrations | Baseline, post treatment (approximately 4 hours)
  Measurement of plasma free fatty acid (FFA) concentrations from femoral, upper body subcutaneous adipose tissue expressed as nmol•million adipocytes-1•min-1

SECONDARY OUTCOMES:
pHSL/HSL response | approx. 6 hours
  Measure of pHSL/HSL level in subcutaneous biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials